CLINICAL TRIAL: NCT00016913
Title: Phase II Study Of Neo-Adjuvant Paclitaxel, Estramustine And Carboplatin (TEC) Plus Androgen Ablation Prior To Radiation Therapy In Patients With Poor Prognosis Localized Prostate Cancer
Brief Title: Chemotherapy, Hormone Therapy, and Radiation Therapy in Treating Patients With Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-99811; U10CA031946 (NIH); CALGB-99811; CDR0000068632 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Carboplatin; Estramustine; Paclitaxel; Radiotherapy; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neo-Adj ChemoTx + ablation prior to RT (Experimental): Patients with localized high-risk prostate cancer were treated with 4 cycles (16 weeks) of continuous weekly paclitaxel at 80 mg/m^2 intravenously with estramustine at 280 mg orally 3 times a day for 5 days a week and carboplatin (area under the curve of 6) on Day 1 of every cycle followed by 3-dimensional conformal or intensity-modulated radiotherapy (total dose of 77.4 gray [Gy] in 1.8-Gy fractions). All patients received androgen deprivation therapy with either goserelin acetate at 3.6 mg subcutaneously or leuprolide acetate at 7.5 mg intramuscularly monthly for 6 months starting at Day 1 of therapy.
  Interventions: Drug: carboplatin; Drug: estramustine; Drug: paclitaxel; Radiation: radiation therapy; Drug: leuprolide or goserelin acetate

INTERVENTIONS:
Drug: carboplatin — AUC=6 week one of each 4 week cycle
Drug: estramustine — 2 tablets tid PO 5 of 7 days per week each 4 week cycle
Drug: paclitaxel — 80 mg/sq m IV infusion over 1 hour weekly for ea 4 week cycle
Radiation: radiation therapy — 77.4 Gy in 1.8 Gy fractions
Drug: leuprolide or goserelin acetate — 7.5 mg IM injection once every 4 weeks for 6 months

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Androgens can stimulate the growth of prostate cancer cells. Drugs such as goserelin or leuprolide may stop the adrenal glands from producing androgens. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy, hormone therapy, and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying giving chemotherapy together with hormone therapy and radiation therapy in treating patients with locally advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and safety of paclitaxel, estramustine, carboplatin, and androgen ablation followed by radiotherapy in patients with poor-prognosis locally advanced prostate cancer.
* Determine the progression-free survival and time to prostate specific antigen failure in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 1 hour once weekly; oral estramustine three times a day, five days a week; and carboplatin IV over 1 hour once monthly. Treatment repeats every 4 weeks for 4 courses.

Patients also receive gonadotropin-releasing hormonal therapy comprising either goserelin subcutaneously or leuprolide intramuscularly once monthly. Treatment repeats every 4 weeks for 6 courses.

After the completion of chemotherapy, patients undergo radiotherapy once daily on weeks 17-24.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 1.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate with one of the following prognostic factors:

  * Tx N0, baseline prostate specific antigen (PSA) greater than 20 ng/mL, and Gleason score at least 7
  * T3b-4 N0, any baseline PSA, and any Gleason score
* No pelvic lymph node disease requiring pelvic radiotherapy
* No metastatic disease by bone scan, CT scan, or MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 1.5 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* No significant cardiovascular disease
* No New York Heart Association class III or IV congestive heart failure
* No active angina pectoris
* No myocardial infarction within the past 6 months
* No history of hemorrhagic or thrombotic cerebral vascular accident
* No deep vein thrombosis within the past 6 months

Pulmonary:

* No pulmonary embolism within the past 6 months

Other:

* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for prostate cancer
* No concurrent routine filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy:

* No prior chemotherapy for prostate cancer
* No other concurrent anticancer chemotherapy

Endocrine therapy:

* No more than 6 weeks of prior androgen deprivation therapy
* No other concurrent anticancer hormonal therapy except steroids for adrenal failure and/or hormones for nondisease-related conditions (e.g., insulin for diabetes)

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy for prostate cancer
* No other concurrent anticancer radiotherapy

Surgery:

* At least 4 weeks since prior major surgery

Other:

* No prior alternative therapy (e.g., PC-SPES) for prostate cancer
* No concurrent alternative medicine (e.g., PC-SPES or saw palmetto) or large quantities of vitamins
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2001-05; Primary Completion 2007-07 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William K. Kelly, DO, Study Chair — Yale University
Locations (23):
- United States (23):
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Veterans Affairs Medical Center - Baltimore, Baltimore, Maryland
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oswego Hospital, Oswego, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Community General Hospital of Greater Syracuse, Syracuse, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Danville Regional Medical Center, Danville, Virginia

REFERENCES:
- [Result] Kelly WK, Halabi S, Elfiky A, Ou SS, Bogart J, Zelefsky M, Small E; Cancer Leukemia Group B. Multicenter phase 2 study of neoadjuvant paclitaxel, estramustine phosphate, and carboplatin plus androgen deprivation before radiation therapy in patients with unfavorable-risk localized prostate cancer: results of Cancer and Leukemia Group B 99811. Cancer. 2008 Dec 1;113(11):3137-45. doi: 10.1002/cncr.23910. PMID 18989865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 15, 2001 and June 30, 2006, a total of 34 patients were enrolled in the study. All CALGB institutions, comprised of 29 major university medical centers and their affiliates, were approved to participate in this study, of which 10 CALGB sites enrolled patients.
Pre-assignment Details: Of these 34 patients, 4 patients did not have radiotherapy, 2 patients were ineligible, and 1 case had limited follow-up data after radiotherapy. Final analyses were performed on 27 patients.
Groups:
- Neo-Adj ChemoTx + Ablation Prior to RT: Treatment with chemotherapy plus androgen ablation prior to radiation treatment for poor prognosis localized prostate cancer
Period: Overall Study
Arm/Group | Neo-Adj ChemoTx + Ablation Prior to RT
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neo-Adj ChemoTx + Ablation Prior to RT
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 61 [52 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Toxicity
Description: Patients were evaluated for acute toxicities defined as grade 3 or greater cardiovascular (including venous thrombosis), gastrointestinal, or genitourinary toxicity occurring during the period starting from treatment initiation until 90 days or less after the completion of radiotherapy. The same toxicity measures were monitored at >90 days after the completion of radiotherapy.
Time Frame: 90 days and 1 year post treatment
Population: Final analyses were performed on all 27 eligible patients.
Measure: Number; unit: Events
Arm/Group | Neo-Adj ChemoTx + Ablation Prior to RT
Number analyzed (Participants) | 27
Events
  Grade 3+ Toxicity <=90 days post radiotherapy | 2
  Grade 3+ Toxicity >90 days post radiotherapy | 0

2. Secondary Outcome: Time to Prostate-specific Antigen Failure
Description: PSA progression was defined in 2 ways. The CALGB PSA progression was defined as 2 consecutive rises in PSA with a rise of at least 0.2 ng/mL and above 1.0 ng/mL after radiation therapy; the date of PSA failure is taken as the midpoint between the last PSA before the rise and the first of the 2 PSAs that documented the rise. In addition, PSA progression was used according to the American Society for Therapeutic Radiology and Oncology 1996 (ASTRO) criteria and defined as 3 consecutive rises in PSA after radiation therapy. The date of PSA failure was taken as the midpoint between the time of the lowest PSA measure after irradiation and the first of the 3 consecutive rises.
Time Frame: PSA was measured every 4 weeks during chemotherapy, at least every 12 weeks post radiation for 2 years, and every 6 months thereafter until PSA failure date (Up to 5.5 years).
Population: All 27 evaluable patients were used in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neo-Adj ChemoTx + Ablation Prior to RT
Number analyzed (Participants) | 27
months
  CALGB criteria | 17.1 [13.3 to 25.9]
  ASTRO criteria | 12.1 [10.3 to 15.7]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time between treatment initiation and the date of disease progression (PSA, bone, tumor) or death, whichever occurred first. PSA progression is defined as 2 consecutive rising PSAs (a rise of at least 0.2 ng/mL) above 1.0 ng/mL.
Time Frame: registration to progression, up to 5.5 years from registration
Population: All 27 evaluable patients were used in this analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Neo-Adj ChemoTx + Ablation Prior to RT
Number analyzed (Participants) | 27
months | 12.1 [10.3 to 15.7]

ADVERSE EVENTS:
Description: All patients that received protocol treatment were analyzed for Adverse Events. Of the 34 patients that enrolled, 4 patients did not have radiotherapy and 1 patient was not evaluated for adverse events. Therefore, 29 patients were evaluated for adverse events.
Arm/Group | Neo-Adj ChemoTx + Ablation Prior to RT
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 29/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neo-Adj ChemoTx + Ablation Prior to RT (N=29)
Blood disorder (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 27 (106)
Hemolysis (Blood and lymphatic system disorders) | 2 (3)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 2 (2)
Edema (Cardiac disorders) | 14 (31)
Left ventricular failure (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Endocrine disorder (Endocrine disorders) | 3 (4)
Diplopia (Eye disorders) | 1 (1)
Eye disorder (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (9)
Constipation (Gastrointestinal disorders) | 18 (27)
Diarrhea (Gastrointestinal disorders) | 17 (36)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 2 (3)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 17 (29)
Proctitis (Gastrointestinal disorders) | 6 (9)
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 7 (9)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3)
Rectal pain (Gastrointestinal disorders) | 6 (12)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (9)
Chest pain (General disorders) | 2 (4)
Fatigue (General disorders) | 25 (102)
Fever (General disorders) | 4 (4)
General symptom (General disorders) | 1 (1)
Ill-defined disorder (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 8 (21)
Radiation-Other(Specify,_____) (General disorders) | 1 (1) — Swelling
Catheter related infection (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 8 (10)
Nail infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urethral infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 9 (9)
Alanine aminotransferase increased (Investigations) | 11 (15)
Alkaline phosphatase (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 9 (22)
Blood bilirubin increased (Investigations) | 5 (6)
Coagulopathy (Investigations) | 1 (1)
Creatine phosphokinase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 13 (24)
Forced expiratory volume decreased (Investigations) | 1 (1)
INR increased (Investigations) | 15 (17)
Laboratory test abnormal (Investigations) | 1 (4)
Leukocyte count decreased (Investigations) | 18 (58)
Lymphocyte count decreased (Investigations) | 9 (35)
Neutrophil count decreased (Investigations) | 10 (12)
Platelet count decreased (Investigations) | 15 (34)
Serum cholesterol increased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (2)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (10)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 23 (71)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 10 (23)
Serum calcium decreased (Metabolism and nutrition disorders) | 14 (29)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 3 (5)
Serum phosphate decreased (Metabolism and nutrition disorders) | 5 (6)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (6)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 13 (24)
Serum sodium increased (Metabolism and nutrition disorders) | 2 (2)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (7)
Dysgeusia (Nervous system disorders) | 7 (8)
Extrapyramidal disorder (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 7 (9)
Neuralgia (Nervous system disorders) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 18 (57)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 8 (11)
Libido decreased (Psychiatric disorders) | 3 (4)
Personality change (Psychiatric disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 3 (4)
Dysuria (painful urination) (Renal and urinary disorders) | 14 (30)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 9 (12)
Incontinence (Renal and urinary disorders) | 2 (2)
Ureteric perforation (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 26 (113)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 6 (10)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 4 (5)
Erectile dysfunction (Reproductive system and breast disorders) | 13 (36)
Gynecomastia (Reproductive system and breast disorders) | 5 (16)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Penile pain (Reproductive system and breast disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 14 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (16)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (12)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 3 (3)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 13 (23)
Hypertension (Vascular disorders) | 4 (5)
Hypotension (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No